CLINICAL TRIAL: NCT01210170
Title: Acute Effect of Mometasone Furoate DPI on Beta-adrenergic Airway and Airway Vascular Relaxation in Moderately Severe Asthma
Brief Title: Acute Effect of Mometasone on Beta-adrenergic Airway and Airway Vascular Relaxation in Severe Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Adam Wanner, Professor of Medicine, University of Miami
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 20071188; P05299 (Other: Sponsor)
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-10

CONDITIONS: Asthma
Keywords: asthma,; inhaled corticosteroids,; airway blood flow,; mometasone,; albuterol; spirometry
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- mometasone 400 mcg - 30 min (Experimental): randomly assigned intervention
  Interventions: Drug: mometasone 400 mcg
- mometasone 400 mcg simultaneous (Experimental): randomly assigned intervention
  Interventions: Drug: mometasone 400 mcg
- placebo- 30 min (Placebo Comparator): randomly assigned intervention
  Interventions: Drug: placebo
- placebo simultaneous (Placebo Comparator): randomly assigned intervention
  Interventions: Drug: placebo
- mometasone 400 mcg - 60 min (Experimental): randomly assigned intervention
  Interventions: Drug: mometasone 400 mcg
- placebo- 60 min (Placebo Comparator): randomly assigned intervention
  Interventions: Drug: placebo
- mometasone 200 mcg - 30 min (Experimental): randomly assigned intervention
  Interventions: Drug: mometasone 200 mcg
- mometasone 200 mcg - 60 min (Experimental): randomly assigned intervention
  Interventions: Drug: mometasone 200 mcg
- mometasone 200 mcg simultaneous (Experimental): randomly assigned intervention
  Interventions: Drug: mometasone 200 mcg

INTERVENTIONS:
Drug: placebo — placebo inhalation before albuterol.
  Other Names: Asmanex placebo
  Arms: placebo simultaneous; placebo- 30 min; placebo- 60 min
Drug: mometasone 400 mcg — mometasone inhalation before albuterol.
  Other Names: Asmanex
  Arms: mometasone 400 mcg - 30 min; mometasone 400 mcg - 60 min; mometasone 400 mcg simultaneous
Drug: mometasone 200 mcg — 200ug mometasone before albuterol.
  Other Names: Asmanex
  Arms: mometasone 200 mcg - 30 min; mometasone 200 mcg - 60 min; mometasone 200 mcg simultaneous

SUMMARY:
Glucocorticosteroids inhibit the disposal of organic cations by blocking organic cation transporters expressed by non-neuronal cells, thereby interfering with the inactivation of the organic cations by intracellular enzymes. Beta2-adrenergic agonists are organic cations, and the concentration of inhaled beta2-adrenergic agonists at beta2-adrenergic receptor sites on smooth muscle is likely to be increased by inhaled glucocorticosteroids (ICS) by the ICS' effect on the glucocorticosteroid-sensitive organic cation transporters. The investigators have shown in human airway vascular smooth muscle cells that the glucocorticosteroid action on organic cation uptake occurs within minutes, does not involve gene transcription or protein synthesis, is not mediated through classical steroid receptors, and is cell membrane-linked.

In the present proposal, the investigators wish to use different single doses of mometasone, a clinically effective ICS, administered with or at different times before albuterol inhalation in subjects with moderate persistent asthma who are obstructed at the time of study.

With this approach the investigators will test the hypothesis that a single inhalation of mometasone causes an acute, transient, dose-dependent potentiation of beta2-adrenergic bronchodilation.

If the hypothesis that a single dose of mometasone acutely potentiates beta2-adrenergic bronchodilation is correct, the results would have a significant impact on treatment strategies involving ICSs and beta2-adrenergic agonists in patients with asthma.

DETAILED DESCRIPTION:
Fifteen non-smokers (males and females between the ages of 18 and 65 years) with physician-diagnosed moderate persistent asthma will be recruited for the study. The subjects will be allowed to use inhaled controller (including ICS) and rescue medication. At study entry, all asthmatic subjects must be clinically stable, and have a forced pre-bronchodilator one-second expired volume (FEV1) of < 75% predicted.

Approval for the protocol will be requested from the University of Miami Institutional Review Board. All subjects will provide written informed consent.

Exclusion criteria:

* Cardiovascular disease and use of cardiovascular medications
* Pregnancy
* Use of oral controller medication for asthma (methylxanthines, systemic glucocorticosteroids, leukotriene modifiers)
* An acute respiratory infection within 4 weeks before enrollment.

Each subject will make 8 visits to the research laboratory.

Procedures:

Visit 1 (screening visit): On this visit, after having signed the consent form, the subjects will perform spirometry before and 15 min after inhaling 180 µg albuterol from a HFA-MDI using a spacer.

Visit 2-8:Subjects that qualify for the study will be asked to return for 7 more visits for the following treatment protocols:

* Inhalation of 400 µg mometasone 30 min before inhalation of 180 µg albuterol
* Inhalation of mometasone placebo 30 min before inhalation of 180 µg albuterol
* Simultaneous inhalation of 400 µg mometasone and 180 µg albuterol
* Simultaneous inhalation of mometasone placebo and 180 µg albuterol

Systemic blood pressure, pulse, O2 saturation, spirometry and airway blood flow ( Qaw) will be measured before mometasone or placebo inhalation, and before and 15 min after albuterol inhalation except on the day when mometasone and albuterol are co-administered; on that day the measurements will be made before and 15 min after the mometasone/albuterol co-administration.

ELIGIBILITY:
Inclusion Criteria:Fifteen non-smokers (males and females between the ages of 18 and 65 years) with physician-diagnosed moderate persistent asthma and FEV1 < 75% of predicted.

Exclusion Criteria:Cardiovascular disease and use of cardiovascular medications, pregnancy, use of oral controller medication for asthma (methylxanthines, systemic glucocorticosteroids, leukotriene modifiers), an acute respiratory infection within 4 weeks before enrollment

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wanner, Principal Investigator — University of Miami
Locations (1):
- Human Research Laboratory- University of Miami School of Medicine, Miami, Florida, United States

REFERENCES:
- [Derived] Mendes ES, Cadet L, Arana J, Wanner A. Acute effect of an inhaled glucocorticosteroid on albuterol-induced bronchodilation in patients with moderately severe asthma. Chest. 2015 Apr;147(4):1037-1042. doi: 10.1378/chest.14-1742. PMID 25611803

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: • Inhalation of 400 µg mometasone DPI 30 min before inhalation of 180 µg albuterol
  Mometasone furoate: • Inhalation of 400 µg mometasone or placebo DPI 30 min before inhalation of 180 µg albuterol
  • Inhalation of 400 µg mometasone or placebo DPI 60 min before inhalation of 180 µg albuterol
Period: Overall Study
Arm/Group | All Study Participants
Started | 22
Completed | 15
Not Completed | 7

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: • participant with asthma were enrolled in the study
Arm/Group | All Study Participants
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Albuterol-induced Change in FEV1
Description: FEV1 will be measured before and after inhalation of 180 mcg albuterol.
Time Frame: 15 minutes after albuterol inhalation
Population: As specified by the protocol, -60 minutes values were not to be analyzed if 200 mcg and 400 mcg of mometasone given 30 minutes before albuterol were determined to have no effect
Measure: Mean (Standard Error); unit: liters
Groups:
- All Participants Received 400 mcg Mometasone-30 Min: mometasone 400 mcg 30 minutes before albuterol 180 mcg inhalation
- All Participants Received Placebo 30 Minutes Before Albuterol: mometasone placebo 30 minutes before albuterol 180 mcg inhalation
- All Participants Received 400 mcg Mometasone Simultaneous: inhalation of 400 mcg mometasone immediately before inhalation of 180 mcg albuterol
- All Participants Received Placebo Simultaneously With Albutero; All Participants Received 200 mcg Mometasone Simultaneous: inhalation of mometasone placebo immediately before inhalation of 180 mcg albuterol.
- All Participants Received 200 mcg Mometasone-30 Min: mometasone 200 mcg 30 minutes before inhalation of 180 mcg of albuterol
- All Participants Received 400 mcg -60 Min: mometasone 400 mcg 60 minutes before inhalation of 180 mcg of albuterol
- All Participants Received Placebo -60 Min: placebo 60 minutes before inhalation of 180 mcg of albuterol
- All Participants Received 200 mcg -60 Min: mometasone 200 mcg 60 minutes before inhalation of 180 mcg of albuterol
Arm/Group | All Participants Received 400 mcg Mometasone-30 Min | All Participants Received Placebo 30 Minutes Before Albuterol | All Participants Received 400 mcg Mometasone Simultaneous | All Participants Received Placebo Simultaneously With Albutero | All Participants Received 200 mcg Mometasone-30 Min | All Participants Received 400 mcg -60 Min | All Participants Received Placebo -60 Min | All Participants Received 200 mcg Mometasone Simultaneous | All Participants Received 200 mcg -60 Min
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15
liters | 0.27 (0.04) | 0.18 (0.04) | 0.32 (0.04) | 0.20 (0.05) | 0.23 (0.04) | NA (NA) — Prespecified data were not analyzed due to the -30min results | NA (NA) — were not analyzed due to the -30min results | NA (NA) — were not analyzed due to the -30min results | NA (NA) — were not analyzed due to the -30min results

2. Secondary Outcome: Albuterol Induced Percent Change in Qaw
Description: Qaw will be measured before and 15 min after albuterol inhalation
Time Frame: change in Qaw 15 minutes after albuterol inhalation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percent change in Qaw
Groups:
- 400 mcg Mometasone 30 Minutes Before Albuterol: • Inhalation of 400 µg mometasone 30 min before inhalation of 180 µg albuterol
- Mometasone Placebo 30 Minutes Before Albuterol: Inhalation of mometasone placebo 30 min before inhalation of 180 µg albuterol
- 400 mcg Mometasone and Albuterol Simultaneously: inhalation of 400 mcg mometasone immediately before inhalation of 180 mcg albuterol.
- Mometasone Placebo and Albuterol Simultaneously: inhalation of mometasone placebo immediately before inhalation of 180 mcg albuterol.
- 400 mcg Mometasone 60 Minutes Before Albuterol: Inhalation of 400 µg mometasone 60 min before inhalation of 180 µg albuterol
- Mometasone Placebo 60 Minutes Before Albuterol: Inhalation of mometasone placebo 60 min before inhalation of 180 µg albuterol
- 200 mcg Mometasone and Albuterol Simultaneously: inhalation of 200 mcg mometasone immediately before inhalation of 180 mcg albuterol
- 200 mcg Mometasone 60 Minutes Before Albuterol: Inhalation of 200 µg mometasone 60 min before inhalation of 180 µg albuterol
- 200 mcg Mometasone 30 Minutes Before Albuterol: Inhalation of 200 µg mometasone 30 min before inhalation of 180 µg albuterol
Arm/Group | 400 mcg Mometasone 30 Minutes Before Albuterol | Mometasone Placebo 30 Minutes Before Albuterol | 400 mcg Mometasone and Albuterol Simultaneously | Mometasone Placebo and Albuterol Simultaneously | 400 mcg Mometasone 60 Minutes Before Albuterol | Mometasone Placebo 60 Minutes Before Albuterol | 200 mcg Mometasone and Albuterol Simultaneously | 200 mcg Mometasone 60 Minutes Before Albuterol | 200 mcg Mometasone 30 Minutes Before Albuterol
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15
percent change in Qaw | 18 (3) | 0 (3) | 30 (7) | -2 (3) | NA (NA) — data not analyzed | NA (NA) — data not analyzed | NA (NA) — data not analyzed | NA (NA) — data not analyzed | NA (NA) — data not analyzed

ADVERSE EVENTS:
Groups:
- All Study Participants: Simultaneous inhalation of 400 µg mometasone DPI and 180 µg albuterol
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes